CLINICAL TRIAL: NCT04357990
Title: Use of a Medical Device, Viruxal Oral and Nasal Spray, for Treating the Symptoms of COVID-19 Via Application to the Naso- and Oropharyngeal Mucosa
Brief Title: Viruxal Oral and Nasal Spray for Treating the Symptoms of COVID-19
Acronym: KONS-COVID19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerecis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS-0470
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Viruxal Oral and Nasal Spray (Experimental): The Device will be administered to the oral and nasal passages, three times per day.
  Interventions: Device: Viruxal Oral and Nasal Spray
- Placebo (Placebo Comparator): The placebo will be administered to the oral and nasal passages, three times per day.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Viruxal Oral and Nasal Spray — Viruxal Oral and Nasal Spray is a Class I CE marked medical device manufactured by Kerecis hf. The Device contains Omega3 Viruxide. The main components in Omega3 Viruxide are Neem oil and St. John's Wort oil. The Device is administered from a pressurized canister into the oral and nasal cavity, where it creates a physical barrier for temporary protection of the mucosal tissue.
  Arms: Viruxal Oral and Nasal Spray
Other: Placebo — The placebo will be a similar spray containing saline only.
  Arms: Placebo

SUMMARY:
Viruxal Oral and Nasal Spray is a Class I CE marked medical device manufactured by Kerecis hf (the "Device"). A double blind clinical trial will be conducted to evaluate the Device against placebo in COVID-19 positive, symptomatic patients in Iceland. Immediate access to COVID-19 patients is available through a well-organized COVID-19 outpatient follow-up clinic. Up to 128 patients with mild to moderate symptoms of COVID-19 will be recruited (so called "higher end of the low risk group"). These patients will be positive for COVID-19, be symptomatic with upper respiratory symptoms, but without involvement of the entire respiratory system. The patients will be randomized to receive treatment with the Study Device or to receive placebo. 64 patients will be randomized into the Study Device group and 64 patients into the Control group. Patients will administer Study Device or Control for 14 days and will have their symptoms recorded until no further symptoms are reported, up to a maximum of 28 days follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Positive for SARS-CoV-2 infection
* Has symptoms of upper respiratory infection
* Willing to participate in the clinical trial and gives consent
* Is not pregnant, nor actively trying to conceive a child.

Exclusion Criteria:

* Under 18 years of age
* Negative for SARS-CoV-2 infection
* Severe symptoms of infection
* Symptoms involving the entire respiratory system, including Pneumonia
* Requires hospitalisation prior to study start
* Asymptomatic
* Pregnant or actively trying to conceive a child
* Other comorbidities that would prevent administration of the device
* Requirement to take regular medications administered by inhalation, or via the naso- and oropharyngeal route
* Patients with known allergies to Neem or Hypericum oil
* Patients with asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Number of days until complete resolution of symptoms per group | 28 days
  The number of days until participants report no symptoms, which they attribute to COVID-19, will be compared between groups. Symptoms include: Fever (38.0°C or higher), chills, dry cough, cough with rise, shortness of breath (rest), shortness of breath (Exercise), dyspnoea, sore throat, runny nose, headache, myalgia/bone pain, anorexia, nausea, vomiting, loss of smell, osteoporosis, abdominal pain, diarrhea, weakness.
Number of hospital admissions per group | 28 days
  The number of participants admitted to hospital due to deterioration of their condition due to COVID-19 will be compared between groups.

SECONDARY OUTCOMES:
Number of days until a reduction in symptoms per group | 28 days
  The number of days until participants report a reduction in symptoms, which they attribute to COVID-19, will be compared between groups.
  Symptoms include: Fever (38.0°C or higher), chills, dry cough, cough with rise, shortness of breath (rest), shortness of breath (Exercise), dyspnoea, sore throat, runny nose, headache, myalgia/bone pain, anorexia, nausea, vomiting, loss of smell, osteoporosis, abdominal pain, diarrhea, weakness.
Number of adverse events per group | 28 days
  The number of adverse events reported will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ragnar F Ingvarsson, MD, Principal Investigator — Landspitalinn University Hospital, Iceland
Locations (1):
- National Hospital of Iceland (Landspítali), Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No